CLINICAL TRIAL: NCT05230784
Title: Effectiveness of Indoor Air Purifiers on Heart Failure Outcomes
Brief Title: The PURI-HF (Air Purifiers on Heart Failure) Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-00954; R01ES033222 (NIH)
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Indoor Air Purifier
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEPA Air Purifier (Experimental): Air purifier is installed in participants' households by the research team. Twice per year, participants will wear a GPS as well as a backpack containing a particulate matter 2.5 (PM2.5) personal exposure monitor for a 24-hour monitoring period.
  Interventions: Other: AirOk Air Purifier
- EGAPA Air Purifier (Placebo Comparator): Air purifier is installed in participants' households by the research team. Twice per year, participants will wear a GPS as well as a backpack containing a particulate matter 2.5 (PM2.5) personal exposure monitor for a 24-hour monitoring period.
  Interventions: Other: Placebo Air Filter

INTERVENTIONS:
Other: AirOk Air Purifier — The AirOk purifier nests on a locally developed patented technology that combines HEPA (grade H12) and a novel EGAPA (Effective Granular Adsorbent Particulate Arrestor) to reduce indoor air pollution. The HEPA filter removes all particulate matter up to 0.3 µm in aerodynamic diameter, and the dual stratified EGAPA filter removes other pollutants such as sulfur, nitrous oxide, carbon oxide, volatile organic compounds, allergens, and mold.
  Arms: HEPA Air Purifier
Other: Placebo Air Filter — Participants in the placebo arm will receive an air purifier with only the EGAPA filter.
  Arms: EGAPA Air Purifier

SUMMARY:
Indoor air pollution and fine mode particulate matter with an aerodynamic diameter smaller than 2.5 micrometers (PM2.5) is a major contributor to global morbidity and mortality, particularly due to cardiovascular disease. This project aims to demonstrate the efficacy, feasibility and effectiveness of portable air filters in improving indoor PM2.5 levels and improving functional capacity of heart failure patients with reduced ejection fraction in India. The findings from the project will add to existing knowledge of innovative and scalable strategies to improve environmental and cardiovascular health worldwide.

The overall objective of this study is to demonstrate the efficacy, feasibility, and effectiveness of portable air filters in improving indoor PM2.5 levels and improving functional capacity of heart failure patients with reduced ejection fraction in India.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age diagnosed with HF with a reduced ejection fraction of ≤ 40% within the last six months in NYHA class II-IV.

Exclusion Criteria:

* listed for a cardiac transplant
* history of CRT device implantation in last 3 months
* on oxygen therapy
* with severe pulmonary disease
* participants unable to ambulate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Distance Walked | Baseline, 12 months
  The distance in meters will be recorded during a 6-minute walk test (MWT)

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) | Baseline, 12 months
Change in Diastolic Blood Pressure (DBP) | Baseline, 12 months
Change in Heart Rate | Baseline, 12 months
Change in pro B-type natriuretic peptide (Pro-BNP) Levels | Baseline, 12 months
Change in Number of Hospitalizations | Baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Vedanthan, MD, MPH, Principal Investigator — NYU Langone Health
Locations (3):
- India (3):
  - Centre for Chronic Disease Control (CCDC), Thiruvananthapuram, Kerala
  - All India Institute of Medical Sciences (AIIMS), Delhi, Punjab
  - Public Health Foundation of India (PHFI), Ludhiana, Punjab

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access upon reasonable request. Requests should be directed to rajesh.vedanthan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.